CLINICAL TRIAL: NCT00111943
Title: Phase II Expanded Safety and Acceptability Study of the Vaginal Microbicide 1% Tenofovir Gel
Brief Title: Safety and Acceptability of a Vaginal Microbicide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HPTN 059; 10145 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hepatitis B, Chronic
Keywords: Anti-Infective Agents, Local; HIV Seronegativity; Tenofovir; Vaginal gel; Microbicide; Vaginal Microbicide; PMPA
MeSH Terms: conditions — HIV Infections; Hepatitis B, Chronic

INTERVENTIONS:
Drug: 1% tenofovir gel

SUMMARY:
The purpose of this study is to determine the safety and acceptability of a vaginal microbicide in HIV uninfected sexually active women.

Study hypothesis: The vaginal microbicide 1% tenofovir will be safe and well tolerated in HIV uninfected women who are in good general health.

DETAILED DESCRIPTION:
While the male condom is effective in preventing sexual transmission of HIV, its use is hampered by deeply rooted cultural and social barriers. About half of all HIV infections worldwide occur in women, yet the only available female-controlled method of HIV prevention is the female condom. Alternative prevention tools, such as vaginal microbicides, are urgently needed to slow the rapid spread of heterosexual HIV infection.

This study will last 24 weeks, with an additional 10 weeks of follow-up for participants with chronic hepatitis B virus (HBV) infection. Participants will be randomly assigned to one of four arms. Arm A participants will insert a vaginal tenofovir 1% gel two hours prior to vaginal intercourse for a maximum of two daily applications. Arm B participants will insert a vaginal placebo gel two hours prior to vaginal intercourse for a maximum of two daily applications. Arm C participants will insert a vaginal tenofovir 1% gel once daily at bedtime or during the longest period of daily rest. Arm D participants will insert a vaginal placebo gel once daily at bedtime or during the longest period of daily rest.

A medical and menstrual history update, pregnancy test, HIV and sexually transmitted infections (STI) risk reduction counseling, and interview to assess behaviors toward vaginal gel use will occur during all study visits. HIV/STI counseling and testing, urinalysis, and blood collection will occur at study entry and at Week 24. Pelvic exam with colposcopy and vaginal swab collection will occur at study entry and Weeks 4, 12, and 24. For participants with chronic HBV, additional blood will be collected to monitor hepatitis B infection at study entry and Weeks 12, 24, 28, 32, and 36.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Good general health
* Sexually active
* Willing to use acceptable methods of contraception, including male latex condoms for all acts of intercourse
* Willing to undergo all study-related assessments and adhere to the requirements of the study

Exclusion Criteria:

* Menopausal or postmenopausal
* Hysterectomy
* Abnormal screening results for several gynecologic exams
* Taking or planning to take tenofovir, adefovir, or any other medication for chronic HBV infection
* History of latex allergy
* History of adverse reaction to tenofovir or adefovir
* Use of a diaphragm or spermicide for contraception
* Prior participation in the study
* Prior participation in any vaginal microbicide, spermicide, or other drug study within 30 days of study entry
* Gynecologic surgical procedure within 90 days of study entry
* Illicit injection drug use within 12 months of study entry
* History of vaginal intercourse more than an average of two times per day in the two weeks prior to study screening
* Any other criteria that, in the investigator's opinion, may interfere with the study
* Current pregnancy or previous pregnancy within 90 days of study entry
* Breastfeeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Macroscopic evidence of damage to the cervical, vulvar, or vaginal epithelium, including ulceration and other lesions, severe erythema, or severe edema, related or not related to the study gel or applicator

SECONDARY OUTCOMES:
Adherence to the study gel regimen
acceptability of the study gel

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hillier, PhD, Study Chair — Department of Obstetrics and Gynecology and Reproductive Sciences, Magee-Women's Hospital; Jessica Justman, MD, Study Chair — Bronx-Lebanon Hospital Center; Smita N. Joshi, MBBS, Study Chair — National AIDS Research Institute (NARI); Craig Hoesley, MD, Study Chair — University of Alabama at Birmingham
Locations (3):
- United States (2):
  - Alabama Microbicide CRS, Birmingham, Alabama
  - Bronx- Lebanon Hospital Center Clinical Research Site (BLHC CRS), The Bronx, New York
- NARI Arogya Aadhar Clinic CRS, Pune, Maharashtra, India

REFERENCES:
- [Background] Bentley ME, Fullem AM, Tolley EE, Kelly CW, Jogelkar N, Srirak N, Mwafulirwa L, Khumalo-Sakutukwa G, Celentano DD. Acceptability of a microbicide among women and their partners in a 4-country phase I trial. Am J Public Health. 2004 Jul;94(7):1159-64. doi: 10.2105/ajph.94.7.1159. PMID 15226137
- [Background] D'Cruz OJ, Uckun FM. Clinical development of microbicides for the prevention of HIV infection. Curr Pharm Des. 2004;10(3):315-36. doi: 10.2174/1381612043386374. PMID 14754390
- [Background] Mantell JE, Myer L, Carballo-Dieguez A, Stein Z, Ramjee G, Morar NS, Harrison PF. Microbicide acceptability research: current approaches and future directions. Soc Sci Med. 2005 Jan;60(2):319-30. doi: 10.1016/j.socscimed.2004.05.011. PMID 15522488
- [Background] Mayer KH, Maslankowski LA, Gai F, El-Sadr WM, Justman J, Kwiecien A, Masse B, Eshleman SH, Hendrix C, Morrow K, Rooney JF, Soto-Torres L; HPTN 050 Protocol Team. Safety and tolerability of tenofovir vaginal gel in abstinent and sexually active HIV-infected and uninfected women. AIDS. 2006 Feb 28;20(4):543-51. doi: 10.1097/01.aids.0000210608.70762.c3. PMID 16470118
- [Background] Van Damme L. Clinical microbicide research: an overview. Trop Med Int Health. 2004 Dec;9(12):1290-6. doi: 10.1111/j.1365-3156.2004.01338.x. PMID 15598260
- See also: Click here for the Alliance for Microbicide Development Web site — http://www.microbicide.org/